CLINICAL TRIAL: NCT04785547
Title: A Phase II Study of Blincyto in Children With CD19+ Precursor B-lineage ALL and MRD-Positivity Before and/or Following First Allogeneic HSCT
Brief Title: ALL SCTped 2012 FORUM Add-on Study Blina Post HSCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by Amgen Limited
Sponsor: Prof. Christina Peters (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Prof. Christina Peters, Univ.-Prof. Dr. Christina Peters, St. Anna Kinderkrebsforschung
Organization: St. Anna Kinderkrebsforschung (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FORUM Add-on Blina post TX
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: ALL, Childhood; Minimal Residual Disease
Keywords: MRD Positivity
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — blinatumomab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Blincyto (Experimental): Blincyto is given over a 28-day cycle. Starting day for patients, who are MRD-positive before HSCT is between day +60 and day +100 and for patients, who become MRD-positive post HSCT it is between day +60 and day +360 post HSCT.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — 15 mcg/m2/day for 28 days
  Other Names: Blincyto

SUMMARY:
An add-on phase II trial within the ALL SCTped 2012 FORUM with the primary objective to determine whether the use of Blincyto in paediatric patients with B-lineage ALL and pre- and/or post-transplant MRD could induce MRD-negativity in patients who were MRD-positive before and/or after allogeneic HSCT.

The study protocol entitled "A Phase II Study of Blincyto (Blinatumomab) in Children with CD19+ B-lineage Acute Lymphoblastic Leukemia (ALL) and Minimal Residual Disease (MRD)-Positivity before or following first Allogeneic Hematopoetic Stem Cell Transplantation (HSCT) in complete remission (CR1, CR2, CR3)" was included in the ALL SCTped 2012 FORUM Protocol Appendix 1b.

According to protocol, 15 mcg/m2/day of Blincyto is given in continuous intravenous infusion over a 28-day cycle. Starting day for patients who are MRD-positive before HSCT is between day +60 and day +100 and for patients who become MRD-positive post HSCT it is between day +60 and day +360 post HSCT.

Patients are evaluated for response at day +28 (+4 days) (bone marrow morphology and MRD analysis - defined by PCR/FLOW-techniques) after start of Blincyto-treatment at the end of first Blincyto infusion and at regular post-TX-checks (according to FORUM: days +28, +60, +100, +180 and +360 after HSCT).

The protocol was approved in 10 countries (Austria, Belgium, Czech Republic, Denmark, France, Italy, Norway, Poland, Slovakia and Spain) participating ALL SCTped 2012 FORUM study. Overall, 3 patients were treated with Blincyto (2 in Oslo and 1 in Copenhagen).

However, the Investigator Initiated Research Agreement was terminated by Amgen on 26 April 2022, leading to an early termination of the study, which was approved with the last protocol amendment.

DETAILED DESCRIPTION:
6.2.1 Screening / Pretreatment* The screening process begins on the date the subject (or legally acceptable representative) signs the IRB/EC approved ICF and assent form and continues until enrollment. Informed consent and assent must be obtained before completing any study-specific procedures. After written informed consent and assent have been obtained, subjects will be screened in order to assess eligibility for study participation. Only eligible subjects who meet the inclusion/exclusion criteria listed in Section 4 will be enrolled in the study. The total screening window is up to 14 days. If a subject has not met all eligibility criteria at the end of the 14-day window, the subject will be classified as a screen failure on the subject screening log. Subjects who screen fail may be eligible to rescreen one time per Section 6.2.2.

The following assessments/procedures are to be completed during the screening period at time points designated in the Schedule of Assessments:

* Confirmation that the Informed Consent Form and Assent Form have been signed
* Product History Form for subjects who were enrolled in a previous Amgen Blincyto study
* Relevant medical history: including all data which are documented in FORUM trial
* Review of inclusion/exclusion criteria
* Physical examination
* Local laboratory assessments within 7 days prior to treatment start:
* Chemistry
* Coagulation
* Hematology (CBC with differential)
* Bone marrow aspirate (morphological and MRD assessment)

  · Lumbar puncture
* Serious Adverse Event reporting 6.2.2 Rescreening* Subjects who are unable to complete or meet eligibility at the initial screening will be permitted to rescreen once, provided study recruitment has not closed. Upon signing a new Informed Consent Form and Assent Form, a new 14-day screening window will begin. Subjects will retain the same subject identification number assigned at the original screening.

After reconsenting, all screening procedures, including the bone marrow aspirate, must be repeated. However, previous bone marrow aspirate/biopsy taken within 14 days of the planned treatment start of Blincyto can be used to determine eligibility.

6.2.3 Treatment* The following procedures will be completed during day 1 to day 29 at the times designated in the Schedule of Assessments. For assessments performed at day 1, all study procedures should be completed prior to the initiation of Blincyto therapy, unless noted otherwise.

* Physical examination (D1 of each treatment cycle), prior to infusion start
* Bone marrow aspirate/biopsy (morphological and MRD assessment): day 29, not mandatory in case of documented disease progression or relapse
* Chemistry, Coagulation, Hematology (Complete blood test (CBC) with differential)
* day 1: +6h after the first dose of Blincyto
* day 2: any time
* day 3: any time
* In addition, hematology only: day 29, not mandatory in case of documented disease progression or relapse.
* Immunoglobulins (IgG only)
* Day 1, prior to infusion start
* Day 29, after end of infusion
* Vital signs (pulse and temperature only), at the following time points:
* Day 1, prior to infusion start
* Day 15 and day 29 (any time)
* Any other time as deemed necessary by the investigator per institutional guidelines
* Neurological examination (eg, finger-nose and/or writing test, as appropriate for age):
* day 1, prior to infusion start
* day 2 and day 3, any time
* Any other time as deemed necessary by the investigator per institutional guidelines
* Serious Adverse Event reporting 6.2.4 Safety Follow-up Visit(s) / End of Study Visit

All subjects, including subjects who withdraw early, should complete a safety follow-up visit 30 days (± 4 days) after the last dose of Blincyto. The following procedures will be completed at the visit:

* Physical examination
* Local laboratory assessments:
* Chemistry
* Coagulation
* Hematology (CBC with differential)
* Immunoglobulins (IgG only)
* Urine or serum pregnancy test (female adolescents of childbearing potential only), if applicable
* Serious Adverse Event reporting 6.2.5 Long-term Follow-up All subjects will be followed in the long-term follow-up portion of the study for OS.

Subjects in remission will also be followed for duration of response. Following the safety follow-up visit, subjects will be followed every 6 months (± 2 weeks) until 14 months after the first dose of Blincyto to assess disease status. The following procedures will be completed for subjects who remain in remission:

* Disease/Survival status
* Bone marrow aspirate/biopsy (morphological and MRD assessment) at day +180 post HSCT and day 360 post HSCT.
* Hematology (neutrophils and platelets) 6.2.6 Lumbar Puncture to Examine Cerebrospinal Fluid In case of clinical signs of CNS-disease a lumbar puncture will be performed as outlined in the Schedule of Assessments to assess for possible leukemic involvement of the CNS. CSF cell count, glucose, and protein will be measured at the local laboratory as part of the examination. Additional investigations of the CSF should be performed as clinically appropriate.

If an Ommaya reservoir is in place and there is no evidence of blockage of CSF flow in the spinal canal, withdrawal of a sample through the Ommaya reservoir is permitted.

6.2.7 Bone Marrow Biopsy / Aspiration

Bone marrow will be used for hematological assessment and for evaluation of MRD. The following samples will be obtained for cytomorphological assessment and MRD measurement by a local laboratory:

* Cytomorphology/percentage of blasts: bone marrow aspirates at screening, at the end of each treatment cycle, and every 6 months during long-term follow-up for subjects in remission only, until relapse.
* MRD: Aliquots at screening will be collected and analyzed. Aliquots for each subsequent bone marrow assessment may be collected and analyzed, if applicable.

In case of insufficient quality of the bone marrow material at the end of each treatment cycle, a repeat bone marrow assessment should be performed prior to treatment start in the next cycle or at the safety follow-up visit if the subject has not progressed and no further treatment cycles are to be administered.

The degree of bone marrow infiltration defined by the percentage of leukemic blasts in bone marrow will be evaluated by local laboratories per cytomorphology and flow cytometry immunophenotyping. During screening the B-precursor phenotype with CD19 positivity (at least partial) should be confirmed for inclusion.

6.2.8 Laboratory Assessments* The analytes for all laboratory tests used throughout this study are listed in the table below. All screening and on-study laboratory samples will be collected and processed at the investigator's local laboratory and analyzed locally. Standard laboratory tests will be performed according to institutional guidelines. The date and time of sample collection will be recorded in the source documents at the site. Blood draws should not be done via the central venous access. Exception: If a permanent central line with more than one lumen is used, blood draws can be done via the lumen that is not used for drug administration. Any additional follow-up laboratory testing should be performed per standard of care for the treatment of ALL and according to ALL SCTped 2012 FORUM-study.

*Numeration as per protocol

ELIGIBILITY:
Inclusion Criteria:

* Patients participating in ALL SCTped 2012 FORUM;
* Age: > 0.5 years and < 21 years;
* B-precursor ALL with < 5% blasts in the bone marrow (M1 bone marrow) and CD19+ minimal residual disease (MRD) before and/or following allogeneic HSCT;
* Indication for first allogeneic HSCT was CD19+ ALL in first, second or third remission;
* Allogeneic Hematopoietic Stem Cell Transplant (HSCT): at first dose of Blincyto patients must be at least > 60 days post-SCT and without evidence of grade 2 or higher acute GVHD and off systemic immunosuppression (tapering allowed) and at least 4 weeks after last donor lymphocyte infusion (DLI);
* Performance-Status (Karnovsky/Lansky): above 50%;
* Written consent of the parents/legal guardian and, if necessary, the minor patient via "Informed Consent Form";
* No pregnancy;
* No secondary malignancy.

Exclusion Criteria:

* Patients who do not fulfill the inclusion criteria;
* The whole protocol or essential parts are declined either by patient himself/herself or the respective legal guardian;
* Malformation syndromes;
* Renal impairment (< 30% of normal glomerular filtration rate);
* Severe pulmonary, hepatic or cardiac impairment due to toxicity or infection (> CTCAE grade 3);
* Recent episode of seizures or posterior reversible encephalopathy syndrome in the past 30 days;

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2022-01-22 (Actual)

PRIMARY OUTCOMES:
Rate of MRD-negativity | Patients may receive 2 cycles of treatment. A single cycle of treatment is 28 days (4 weeks) of continuous infusion. Each cycle of treatment is separated by a 14 day (2 weeks) treatment-free interval.
  Rate of MRD-negativity is defined as < 0.01 percent (%) by flow cytometry and < 10-4 by PCR after first and second Blincyto cycle

CONTACTS AND LOCATIONS:
Overall Officials: Christina Peters, MD, Study Chair — St.Anna Kinderspital, Vienna, Austria
Locations (14):
- St. Anna Kinderspital, Vienna, Austria(AUT), Austria
- University Hospital Gasthuisberg (UZ Leuven), Leuven, Belgium
- Motol University Hospital Prague, Prague, Czechia
- Rigshospitalet Copenhagen, Copenhagen, Denmark
- Hôpital Robert Debré, Paris, Paris, France
- Italy (2):
  - Ospedale S. Gerardo Monza, Monza
  - IRCCS Ospedale Pediatrico Bambino Gesù Roma, Roma
- Oslo University Hospital, Oslo, Norway
- Poland (4):
  - Nicolaus Copernicus University Collegium Medicum, Bydgoszcz
  - Lublin, Medical Academy, Lublin
  - University of Medical Sciences Poznan, Poznan
  - Klinika Transplantacji Szpiku, Wroclaw
- University Children's Hospital, Bratislava, Slovakia
- Hospital Universitario Vall d'Hebron, Barcelona, Spain